| Cover | nage |
|-------|------|
| COVE | page |

Official title: eHealth for nicotine addiction: a feasibility study and pilot RCT

NCT number: NA

Document Date: 11 July 2024

Participant Informed Consent Form

Coach-guided remotely delivered motivational interviewing and cognitivebehavioural therapy for nicotine use disorder: protocol for a feasibility and pilot study

INFORMED CONSENT FORM

(to be completed after the Participant Information Sheet has been read)

**Taking Part** 

Please write your initial to confirm agreement

The purpose and details of this study have been explained to me. I understand that this study is designed to further scientific knowledge and that all procedures have been approved by the Ethics Board (Human Participants) Sub-Committee.

I have read and understood the information sheet and this consent form.

I understand that this programme is not intended to be a first-line treatment for nicotine-related diseases, such as cardiovascular or pulmonary conditions.

I have had an opportunity to ask questions about my participation.

I understand that participating in the study will involve audio recording my feedback on the study or intervention.

I understand that taking part in the study will involve committing to 6 sessions of online treatment for nicotine use disorder.

I understand that the personal information collected will include name, gender, age, ethnicity, and place of residency.

I understand that sensitive personal information including mental health condition, record of health conditions/disabilities, and record of substance misuse, will be collected during this study.

I understand that I am under no obligation to take part in the study, have the right to withdraw from this study at any stage for any reason, and will not be required to explain my reasons for withdrawing.

I understand that I can contact the researcher(s) for this project; by e-mail to receive more information and/or a summary of the anonymised group results.

## Use of Information

I understand that all the personal information I provide will be processed in accordance with data protection legislation on the public task basis and will be treated in strict confidence unless (under the statutory obligations of the agencies which the researchers are working with), it is judged that confidentiality will have to be breached for the safety of the participant or others or for audit by regulatory authorities.

I understand that information I provide will be used for research outputs.

I understand that personal information collected about me that can identify me, such as my name, will not be shared beyond the study team.

I agree that information I provide can be quoted anonymously in research outputs.

If written information is provided by the participant (e.g. diary), I agree to joint copyright of the qualitative data to Overcome.

I understand that anonymised data will be made publicly available on data archiving sites for the purposes of secondary analyses

I understand that this consent form with my name is being collected for the sole purpose of recording that I have agreed to take part and that it will be stored for up to 5 years in Overcome archiving facilities/password protected computer in accordance with relevant data protection policies and regulations, and will be destroyed after 5 years, and no identifying information will be archived for future research and plagiarism checking with the write-up of this project

| Consent to Participate |
|------------------------------------------------|
| I voluntarily agree to take part in this study |
| Name of participant [printed] Signature Date |
| Researcher [printed] Signature Date |
| Researcher [printed] Signature Date |

(Please return this form to this email address: research@overcome.org.uk)